CLINICAL TRIAL: NCT07026981
Title: Exploratory, Prospective, Single-Arm, Open-labeled Study of [Ga68]MTP220 PET for First-in-Human Biodistribution and Efficacy in Patients With Pancreatic Cancer and Head and Neck Cancers
Brief Title: [Ga-68]MTP220 PET for Biodistribution and Efficacy in Pancreatic Cancer and Head and Neck Cancers
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Qiubai Li (Other)
Responsible Party: Sponsor-Investigator, Qiubai Li, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE1Y25
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer; Pancreatic Cancer; Cancer Pancreas
Keywords: [Ga68]MTP220; Positron Emission Tomography Computed Tomography; PET CT Scan
MeSH Terms: conditions — Head and Neck Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [Ga-68]MTP220 PET/CT Imaging (Experimental): Participants will receive an injection of 210 MBq (3.0-6.0 mCi, range 110-220 MBq with an upper limit of 220 MBq) of [Ga68]MTP220 by slow IV push. This will be followed by PET/CT imaging. One diagnostic CT scan will be performed followed by a sequential whole body PET scan (including 7 to 8 fields-of-view depending on participant height) at three points after the injection of the drug. These three points will be 20, 60 and 100 minutes after the injection. Imaging will be performed for about 1 minute per bed position. The total duration of PET data acquisition is about 20-30 minutes.
  Interventions: Drug: [Ga-68]MTP220 PET/CT Scan

INTERVENTIONS:
Drug: [Ga-68]MTP220 PET/CT Scan — Participants will undergo PET/CT imaging after they have received an injection of the targeted PET tracer drug, [Ga-68]MTP220.

SUMMARY:
The goal of this research study is to develop a diagnostic tool to help with detection and diagnosis of head and neck cancer (HNC) and pancreatic cancer (PaC). This tool is called a "targeted PET tracer", or more specifically a drug named "[Ga-68]MTP220". The U.S. Food and Drug Administration (FDA) has not yet approved this drug, so researchers are conducting this research study to see if [Ga-68]MTP220 is safe and effective at diagnosing pancreatic cancer and head and neck cancer. FDA approval has been obtained for this study protocol by an Investigational New Drug (IND) application. Participants will receive a single injection of [Ga-68]MTP220 followed by PET/CT imaging at three points after they received the drug. These study procedures will take about 2.5 hours. Participants will also receive a follow-up phone call the day after receiving the drug to talk about any side effects they experienced.

DETAILED DESCRIPTION:
For HNC, the overall 5-year survival rate of HNSCCs remains ∼40-50%. PaCa is the 3rd leading cause of cancer mortality in the US with its incidence expected to double by 2030. The poor survival of HNC and PaCa patients is partly due to the delayed diagnosis. Thus, early detection and diagnosis is pivotal to improve the survival. Currently, there is still an unmet clinical need for novel diagnostic technologies for early accurate detection and diagnosis of HNC and PaCa. In this exploratory first in human phase 0 trial, researchers are testing the use of a [Ga-68]MTP220 as a targeted PET tracer to explore the biodistribution, dosimetry, efficacy and safety in pancreatic and head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than 18 years old
* Prior biopsy showing pancreatic or head and neck malignancy
* Participants have been newly diagnosed and not yet received definitive therapy (including surgery, radiation therapy, or systemic therapy).
* Able and willing to provide written informed consent before any protocol-specific procedures are undertaken
* Participants willing and able to undergo a PET/CT

Exclusion Criteria:

* Participants who do not meet the above mentioned inclusion criteria
* Participants with severe hepatic and renal dysfunction (Total bilirubin > 3 mg/dL, Albumin < 2.8 g/dL, INR > 2.3 (or prolonged PT), presence of ascites or hepatic encephalopathy (Grade III-IV) End-Stage Renal Disease (ESRD) or eGFR < 30 mL/min/1.73m², Serum creatinine > 4 mg/dL or rapidly rising, Need for dialysis (hemodialysis or peritoneal dialysis), uremic symptoms)
* Participants < 18 years old
* Participants who refuse to give or are unable to sign the informed consent
* Anti-cancer treatment (chemotherapy and/or radiation therapy) within the last 2 weeks
* Participants unable to withstand or undergo PET/CT
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of [Ga-68]MTP220 in patients with pancreatic cancer and head and neck cancers, as measured by standardized uptake value (SUV) mean and maximum | Time it takes to do imaging study procedures, about 2.5 hours
Radiation dosimetry of [Ga-68]MTP220, as measured by dosimetry calculations performed using site software | Time it takes to do imaging study procedures, about 2.5 hours

SECONDARY OUTCOMES:
Safety of [Ga-68]MTP220, as measured by number of participants who experience adverse events (AEs) | Participants will be asked to report AEs via telephone follow-up no more than 1 day after they undergo study imaging
Safety of [Ga-68]MTP220, as measured by number of participants who experience a significant change in blood pressure | Baseline (10 minutes before dose) and at the following points after they received the dose: 10, 50, 90, 140 minutes
  Changes from baseline for vital signs may be tested for differences from zero by time point using ANOVA or paired t-test
Safety of [Ga-68]MTP220, as measured by number of participants who experience a significant change in heart rate | Baseline (10 minutes before dose) and at the following points after they received the dose: 10, 50, 90, 140 minutes
  Changes from baseline for vital signs may be tested for differences from zero by time point using ANOVA or paired t-test
Safety of [Ga-68]MTP220, as measured by number of participants who experience a significant change in respiratory rate | Baseline (10 minutes before dose) and at the following points after they received the dose: 10, 50, 90, 140 minutes
  Changes from baseline for vital signs may be tested for differences from zero by time point using ANOVA or paired t-test
Safety of [Ga-68]MTP220, as measured by number of participants who experience a significant change in blood oxygen saturation | Baseline (10 minutes before dose) and at the following points after they received the dose: 10, 50, 90, 140 minutes
  Changes from baseline for vital signs may be tested for differences from zero by time point using ANOVA or paired t-test
Safety of [Ga-68]MTP220, as measured by number of participants who experience a significant change in electrocardiogram (ECG) | Baseline (10 minutes before dose) and at the following points after the start of they received the dose: 10 and 140 minutes
  Changes in ECG will be summarized using descriptive statistics
Efficacy of [Ga-68]MTP220 PET/CT imaging in detecting PaCa or HNC, as measured by comparison of tumor vs normal tissue uptake of [Ga-68]MTP220, compared to conventional imaging (when available) | Time it takes to do imaging study procedures, about 2.5 hours
  Uptake of [Ga-68]MTP-220 will be assessed by comparing lesion uptake to background activity
Potential of [Ga-68]MTP220 PET/CT for assessing tumor response to immunotherapy in PaCa and HNC, as measured by radiotracer uptake in tumors as compared to background activity, compared to conventional imaging (when available) | Time it takes to do imaging study procedures, about 2.5 hours
  A tumor uptake that is low or approaching background levels-reflected by a low SUVmax is suggestive of a favorable treatment response. In contrast, persistently high uptake may indicate disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Qiubai Li, MD, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No